CLINICAL TRIAL: NCT07238127
Title: Role of AST/ALT Ratio & MPV/Platelets Count Ratio in Breast Cancer
Brief Title: AST/ALT & MPV/Platelets Ratios in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Salah El-Din shaker, Principal investigator, Assiut University
Other Study IDs: AST/ALT & MPV/platelets ratios
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; AST/ALT Ratio; MPV/Platelets Ratio
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims to evaluate the association between AST/ALT ratio and MPV/platelets count ratio with breast cancer in a case-control study.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common malignant tumor in women and the biggest threat to the health of women worldwide. Breast cancer represents a significant global health challenge: it is the most commonly diagnosed cancer in the world with an estimated 2.26 million cases recorded in 2020. Breast cancer is rarely seen in males. The incidence of breast cancer rises rapidly over the years, ranking as the first common cancer among females worldwide, and thus posing a considerable threat to female health. Breast cancer is the leading cause of cancer mortality among females. Although historically considered to be a disease of largely developed countries, over half of breast cancer diagnoses and two-thirds of breast cancer related deaths occurred in the less developed regions of the world in 2020.Being a highly prevalent cancer type, breast cancer is observed in both developing and developed countries with different causes and factors of progression. Adopting new life styles, industrialization, globalization, increased life expectancy, pollution etc are the leading causes of cancer. According to 2018 statistics, every year around 1.2 million new cases of breast cancer were diagnosed. The GLOBACON report of 2018 concluded that breast cancer was the most frequently identified cancer type and leading cause of cancer related death in majority of countries. Major part of breast related cancer is linked with the expression of estrogen receptors and their treatment is related with the disease prognosis. The rate of breast cancer mortality can be reduced down to a limit by early diagnosis; timely treatment and management . The commonly used chemotherapeutic drugs include doxorubicin (DOX), paclitaxel and cyclophosphamide. However, the efficiency of chemotherapy is greatly limited by primary and acquired drug resistance . Chemotherapy is widely accepted as traditional treatment method in spite of the obstacle of chemotherapy resistance. The important mechanisms that may lead to drug resistance include alteration in expression of ABC transporters gene family, damage of topoisomerase enzyme, mutation in DNA repair genes, induced apoptosis by genetic imbalance and alteration in signalling pathways of NF alpha etc. All these worsen the condition of breast cancer making chemotherapy a failure in most cases. According to Yaghoubi et al., 2015, the cells which already acquired drug resistance show cross resistance to anti proliferative nature of anti-oestrogen drugs which have crucial role in breast cancer treatment .

Aspartate aminotransaminase (AST) and alanine aminotransaminase (ALT) are liver enzymes commonly used in clinical laboratory tests. These enzymes released from liver cells into the blood are produced by both malignant and nonmalignant cells.

The AST-ALT ratio, also called the De Ritis ratio, was originally defined by De Ritis in 1957 . Although the De Ritis ratio was first used to identify viral hepatitis and some chronic liver diseases, it has been identified in recent studies as an independent prognostic factor for the prediction of disease stage and patient survival in some malignancies .

Complete blood count (CBC) is a routine test that is frequently requested by physicians to diagnose various diseases, such as anemia, acute infections, bleeding, allergic malignancies, cancers, immune disorder, health screening, and preoperative assessments. It provides critical information about cell types, especially red blood cells (RBC), white blood cells (WBC), and platelets (PLT) . CBC, as a routine and cost-effective test, provides valuable information about various malignancies . Evaluation of the hematological factors is also one of the reliable paraclinical methods to diagnose diseases . Also, hematological parameters have prognosis value in patients with breast cancer . CBC is an essential test for patients with breast cancer before using any treatment .

Thus, considering the importance of hematological parameters in the detection of breast cancer, the aim of this study was to evaluate ALT/AST ratio and MPV/platelets count ratio as useful markers to distinguish between patients with breast cancer and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients of breast cancer admitted to South Egypt Cancer Institute at different stage of the disease

Exclusion Criteria:

1. other malignant diseases
2. male breast cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — females
Study Population: breast cancer patients as cases and healthy people as controls
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Difference in AST/ALT ratio between breast cancer patients and controls 2. Difference in MPV/Platelet count ratio between breast cancer patients and controls | Baseline
  Comparison of mean AST/ALT ratio and MPV/platelets count ratio between the two groups

SECONDARY OUTCOMES:
1. Diagnostic performance of AST/ALT ratio for distinguishing breast cancer patients from controls 2. Diagnostic performance of MPV/Platelet count ratio for distinguishing breast cancer patients from controls | baseline
  Sensitivity, specificity and AUC calculated from AST/ALT ratio and MPV/platelets count ratio values

REFERENCES:
- [Background] Divsalar B, Heydari P, Habibollah G, Tamaddon G. Hematological Parameters Changes in Patients with Breast Cancer. Clin Lab. 2021 Aug 1;67(8). doi: 10.7754/Clin.Lab.2020.201103. PMID 34383417